CLINICAL TRIAL: NCT04782648
Title: Transit Bipartition to Promote Weight Loss After Laparoscopic Sleeve Gastrectomy
Brief Title: Transit Bipartition After Sleeve Gastrectomy
Acronym: TB-LSG
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Markus Reiser, M.D., Chief Dept. Gastroenterology, Ruhr University of Bochum
Other Study IDs: TB-LSG-01
Record Dates: First submitted 2021-02-27; First posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Obesity, Morbid; Weight Gain; Bariatric Surgery Candidate
Keywords: obesity; weight regain; sleeve gastrectomy; SASI bypass
MeSH Terms: conditions — Obesity, Morbid; Weight Gain; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: transit bipartition — transit bipartition as revisional bariatric surgery for weight regain after sleeve gastrectomy
  Other Names: SASI bypass

SUMMARY:
Retrospective analysis of 100 morbidly obese patients who underwent a transit bipartition (TB) procedure ("Single Anastomosis Sleeve Ileal bypass") for inadequate weight loss or weight recidivism after a previous sleeve gastrectomy. Data were collected prospectively in strictly pseudonymous form. The primary endpoint of the study is weight loss at 1, 3, 6 and 12 months after TB. A subgroup analysis evaluates the effect of the length of the common channel. Secondary endpoints include impact on obesity related comorbidities (type 2 diabetes, hypertension, sleep apnea, gastroesophageal reflux) as well as safety.

DETAILED DESCRIPTION:
Prospective data base of 100 consecutive morbidly obese patients who had undergone transit bipartition (TB, also termed "Single Anastomosis Sleeve Ileal bypass") after a previous sleeve gastrectomy (LSG). Inclusion criteria were TB for excess weight loss (EWL) < 50% ≥ 12 months post LSG or weight recidivism of > 5 kg/qm with a body mass index (BMI) > 30 kg/qm. Patients with endocrine disorders other than type 2 diabetes mellitus (T2D), major psychiatric disorders, American Society of Anesthesiologists (ASA) III and higher or pregnant patients were excluded from the study. Data were prospectively collected in strictly pseudonymous form. Follow up time points were at 1, 3, 6 and 12 months following TB. The primary endpoint of the study is weight loss at 1, 3, 6 and 12 months after TB. A subgroup analysis evaluates the effect of the length of the common channel. Secondary endpoints include impact on obesity related comorbidities such as T2D, hypertension, sleep apnea, gastroesophageal reflux as well as safety.

ELIGIBILITY:
Inclusion Criteria:

* TB for excess weight loss (EWL) < 50% ≥ 12 months post LSG or weight recidivism of > 5 kg/qm with a body mass index (BMI) > 30 kg/qm.

Exclusion Criteria:

* endocrine disorders other than T2DM, major psychiatric disorders, ASA ≥ III, pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Morbidly obese patients (BMI > 30) who underwent transit bipartition (SASI bypass) for inadequate weight loss or weight regain after laparoscopic sleeve gastrectomy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
percent excess weight loss (EWL) | 12 months
  preoperative weight-current weight / preoperative weight-ideal weight x 100 (ideal weight defined as BMI 25 kg/qm

SECONDARY OUTCOMES:
number of patients with improvement of type 2 diabetes | 12 months
  number of patients with HbA1c <6 %, fasting blood glucose <100 mg/dL in the absence of antidiabetic medications
number of patients with improvement of gastro-esophageal reflux (GERD) | 12 months
  number of patients with no GERD symptoms, reflux symptom score (RSI) < 13 in the absence of medication
number of patients with improvement of hypertension | 12 months
  number of patients with normotensive blood pressure (<120/80 mmHg) in the absence of antihypertensive medication
number of patients with improvement of sleep apnoea | 12 months
  number of patients with discontinued use of sleep apnea treatment (continuous positive airway pressure - CPAP) based on improved symptoms and Obstructive Sleep Apnoea (OSA) screening.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Reiser, M.D., Principal Investigator — Dept. Gastroenterology, Klinikum-Vest GmbH
Locations (1):
- Klinikum Vest GmbH, Recklinghausen, North Rhine-Westphalia, Germany